CLINICAL TRIAL: NCT04083651
Title: A Phase II/III Adaptive Study to Evaluate the Safety and Efficacy of Oral Methylnaltrexone Bromide Tablets in Subjects With Advanced Pancreatic Cancer
Brief Title: A Study of Methylnaltrexone Bromide (MNTX) in Participants With Advanced Pancreatic Cancer
Status: Withdrawn | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to pandemic challenges and consideration of a different study design in the future.
Sponsor: Bausch Health Americas, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: SAL-REL-2042
Record Dates: First submitted 2019-09-06; First posted 2019-09-10 (Actual); Last update posted 2021-05-07 (Actual); Status verified 2021-05

CONDITIONS: Pancreatic Cancer
MeSH Terms: conditions — Pancreatic Neoplasms | interventions — methylnaltrexone

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Methylnaltrexone Bromide (MNTX) (Experimental): Participants will receive methylnaltrexone bromide (MNTX) 450 mg (3 tablets of 150 mg each) QD orally. If the initial interim analysis suggests a lack of efficacy, subsequent participants will receive 450 mg MNTX twice daily (BID) or three times daily (TID). Treatment will continue until participant's death or early withdrawal from study or study completion at Day 168.
  Interventions: Drug: Methylnaltrexone bromide
- Placebo (Placebo Comparator): Participants will receive placebo matching to MNTX until participant's death or early withdrawal from study or study completion at Day 168.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Methylnaltrexone bromide — Methylnaltrexone bromide will be administered per dose and schedule specified in the respective arm.
  Other Names: Relistor®
  Arms: Methylnaltrexone Bromide (MNTX)
Drug: Placebo — Placebo matching to methylnaltrexone bromide will be administered as mentioned in the respective arm.
  Arms: Placebo

SUMMARY:
This is an adaptive design study. During the first phase of the study, participants will be randomized in 2:1 ratio to receive either MNTX 450 milligrams (mg) once daily (QD) or placebo. An interim analysis will be performed for futility and at that point a higher dosage regimen may be utilized for the active treatment group if the futility criteria are met. For the second stage of the study, interim analyses will be conducted for futility and sample size reassessment.

ELIGIBILITY:
Inclusion Criteria:

* Unresectable adenocarcinoma of the pancreas (other surgery on non-target lesion or unrelated to management of pancreatic adenocarcinoma is not excluded).
* Measurable disease on computed tomography (CT) scan by Response Evaluation Criteria in Solid Tumors (RECIST) 1.1.
* Refused standard chemotherapy, or failed at least one standard of care chemotherapy regimen for pancreatic cancer and refused additional chemotherapy.
* Must be on stable dose of opioids within 2 weeks prior to randomization.
* At least 18 years of age on the date the Informed Consent Form (ICF) is signed and with the capacity to provide voluntary informed consent.
* Must be able to read, understand and provide written informed consent on the Institutional Review Board (IRB)/Ethics Committee (EC) approved ICF and provide authorization as appropriate for local privacy regulations.
* Had no radiotherapy, chemotherapy, or immunotherapy within the 14 days prior to randomization.
* Has no continuing toxicity or potential of delayed toxicity from any prior antineoplastic therapy that can be reasonably anticipated, in the opinion of the principal investigator.
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1, or 2.
* Life expectancy of at least 3 months from date of informed consent.
* Baseline laboratory results as follows: Absolute neutrophil count (ANC) greater than or equal to (≥) 1.0 * 10^9/liter; Platelets ≥50 * 10^9/liter (without platelet transfusion); Bilirubin less than or equal to (≤) 1.5 * upper limit of normal (ULN); Aspartate aminotransferase (AST) ≤5 * ULN; Alanine aminotransferase (ALT) ≤5 * ULN; Negative serum or urine pregnancy test for females of childbearing potential (premenopausal female capable of becoming pregnant).
* Signed an informed consent/Health Insurance Portability and Accountability Act (HIPAA) form.
* Willing and able to comply with scheduled visits, the treatment plan, and laboratory tests.

Exclusion Criteria:

* Concurrent therapy with any other investigational or non-investigational anticancer agent within 14 days of the baseline visit.
* Radiation therapy except for palliative care on a non-target lesion.
* Current use of a peripherally Acting mu-opioid receptor antagonist.
* Be a pregnant or breast-feeding woman.
* Female participants of childbearing potential must agree to use effective contraception method, except if she is of non-childbearing potential, defined as surgically sterile (that is; has undergone complete hysterectomy, bilateral oophorectomy, or tubal ligation at least 3 months earlier) or in a menopausal state (at least 1 year without menses). Male participants must agree to use effective contraception or be surgically sterile (vasectomized for greater than 6 months).
* Have dementia or altered mental status that would prohibit informed consent.
* Diarrhea ≥Grade 1 (Common Terminology Criteria Version 5.0 [CTC V5.0]).
* Bowel obstruction.
* Moderate or severe hepatic impairment (for example; Child-Pugh Class B or C).
* Moderate or severe renal impairment (that is; creatinine clearance less than 60 milliliters/minute as estimated by Cockcroft Gault)
* Have any other unstable medical or psychiatric condition or laboratory abnormality that may increase the risk associated with study participation or study drug administration or may interfere with the interpretation of study results and, in the judgment of the Principal Investigator, would make the participant inappropriate for the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2020-01-06 (Estimated); Primary Completion 2023-10-15 (Estimated); Study Completion 2023-10-15 (Estimated)

PRIMARY OUTCOMES:
Overall Survival | From randomization until death from any cause (up to Day 168)

CONTACTS AND LOCATIONS:
Overall Officials: John Lahey, Study Director — Bausch Health Americas, Inc.
Locations (1):
- Bausch Site 001, Omaha, Nebraska, United States